CLINICAL TRIAL: NCT04678583
Title: Anatomical Resection of Liver MetAstases iN patIents With RAS-mutated Colorectal Cancer
Acronym: ARMANI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VTG-08
Record Dates: First submitted 2020-10-30; First posted 2020-12-22 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Liver Metastasis

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, patient and observer-blinded, confirmatory trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - Anatomical resection (Experimental): removal of the entire, tumor-bearing liver segment(s)
  Interventions: Procedure: Resection of colorectal liver metastases
- B - Non-anatomical resection (Active Comparator): metastasectomy with a margin of healthy liver tissue irrespective of segmental borders
  Interventions: Procedure: Resection of colorectal liver metastases

INTERVENTIONS:
Procedure: Resection of colorectal liver metastases — Comparison of two liver surgery methods

SUMMARY:
the ARMANI trial will test the hypothesis, if an anatomic resection (AR) improves long-term outcome vs. a non-anatomical resection (NAR) in patients undergoing surgery for RAS-mutated colorectal liver metastasis (CRLM).

DETAILED DESCRIPTION:
Despite increasing application and success of personalized treatment in medical oncology, little progress has been made in personalized surgical cancer therapy. The ARMANI trial presents the first prospective, randomized trial to evaluate effectiveness and safety of molecular-guided resection in patients with colorectal liver metastasis (CRLM). While CRLM might be removed independently of the liver's segmental borders, retrospective data favor anatomic resections in the subgroup of patients with a mutation in the RAS oncogene. Therefore, the ARMANI trial will test the hypothesis, if an anatomic resection (AR) improves long-term outcome vs. a non-anatomical resection (NAR) in patients undergoing surgery for RAS-mutated CRLM. The trial will be carried out among 11 high-volume centers of hepato-biliary surgery in Germany. A total of 220 patients will be enrolled and randomized in a 1:1 ratio to undergo an AR vs. NAR. The primary endpoint is intrahepatic disease-free survival (iDFS). In addition, the study will provide important data on perioperative outcomes and quality of life for both surgical techniques. Given the trend among liver surgeons to aim for parenchymal-sparing operations to preserve liver parenchyma, a positive trial will be practice changing and present the first piece of high-level evidence on benefits of personalized surgical therapy guided by the tumor's mutational profile in patients with CRLM.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer with RAS mutation (KRAS or NRAS)
* Colorectal liver metastases (single or multiple)
* Planned R0 resection of liver metastases (and primary tumor, if present)
* Anatomical and non-anatomical liver resection technically feasible
* Male and female patients, age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Extrahepatic metastases
* Planned staged liver resection (e.g. two-stage hepatectomy)
* Diagnosis of another cancer < 5 years prior to randomization Exceptions: curatively treated in situ cervical cancer, curatively resected non-melanoma skin cancer
* Expected lack of compliance
* Addiction or other illnesses which do not allow the person concerned to assess the nature and extent of the clinical trial and its possible consequences

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Intrahepatic disease-free survival (iDFS) | 24 months
  Time from operation date to date of disease recurrence in the liver, followed up at intervals of three months for a maximum duration of 24 months or until death. Any new, solid lesion in the liver after resection of all CRLM that fulfils imaging criteria (CT, MRI) of a metastasis is counted as an iDFS event.

SECONDARY OUTCOMES:
Assessment of additional oncological and perioperative outcomes: Intraoperative blood loss [mL] | During surgery
  Intraoperative blood loss presents the amount of blood lost from skin incision until skin closure. Spilling water and ascites will be subtracted. Swabs will be squeezed and their content will also be sucked and added to the fluid collected in the suction containers.
Assessment of additional oncological and perioperative outcomes: Operating time [min] | During surgery
  Time from skin incision until placement of last skin staple/suture.
Assessment of additional oncological and perioperative outcomes: Transfusion of blood, transfused packed red blood cells (PRBC), fresh frozen plasma (FFP) and / or platelet concentrate (PC) [units] | 48 hours after surgery
  Administration of blood transfusions is documented for the intra- and postoperative period within 48 hours postoperatively.
Assessment of additional oncological and perioperative outcomes: Duration of postoperative hospital stay [days] | At day of discharge, assessed up to 90 days
  Postoperative day 1 until day of discharge
Assessment of additional oncological and perioperative outcomes: Duration of postoperative intermediate/intensive care unit stay [days] | At day of discharge, assessed up to 90 days
  Days on the intermediate care unit (IMC) or intensive care unit (ICU) after surgery. Patient's stay in the recovery room exceeding 24 hours is counted as ICU stay
Assessment of additional oncological and perioperative outcomes: Frequency of peri-operative morbidity after resection | 90 days after surgery
  Frequency of peri-operative complications after resection of the primary tumor
Assessment of additional oncological and perioperative outcomes: Kind of peri-operative morbidity after resection | 90 days after surgery
  Kind of peri-operative complications after resection of the primary tumor
Assessment of additional oncological and perioperative outcomes: 90-day mortality | 90 days after surgery
  Death due to any cause within 90 days after surgery
Assessment of additional oncological and perioperative outcomes: Liver biochemical tests: Platelet count | pre-operatively, 5 days after surgery
  Platelet count will be measured preoperatively and on postoperative day 5
Assessment of additional oncological and perioperative outcomes: Liver biochemical tests: Alanine-aminotransferase | pre-operatively, 5 days after surgery
  Levels of alanine-aminotransferase (ALT) will be measured preoperatively and on postoperative day 5
Assessment of additional oncological and perioperative outcomes: Liver biochemical tests: aspartate-aminotransferase | pre-operatively, 5 days after surgery
  Levels of aspartate-aminotransferase (AST) will be measured preoperatively and on postoperative day 5
Assessment of additional oncological and perioperative outcomes: Liver biochemical tests: Gamma-glutamyl transferase | pre-operatively, 5 days after surgery
  Levels of Gamma-glutamyl transferase (GGT) will be measured preoperatively and on postoperative day 5
Assessment of additional oncological and perioperative outcomes: Liver biochemical tests: International normalized ratio | pre-operatively, 5 days after surgery
  Levels of international normalized ratio (INR) will be measured preoperatively and on postoperative day 5
Assessment of additional oncological and perioperative outcomes: Liver biochemical tests: Total bilirubin | pre-operatively, 5 days after surgery
  Levels of total bilirubin will be measured preoperatively and on postoperative day 5
Assessment of additional oncological and perioperative outcomes: Liver biochemical tests: Albumin | pre-operatively, 5 days after surgery
  Levels of albumin will be measured preoperatively and on postoperative day 5
Assessment of additional oncological and perioperative outcomes: Frequency invasive re-interventions | 30 days after surgery
  Invasive re-interventions such as placement of interventional drains, Endoscopic retrograde cholangiopancreatography (ERCP) with stent placement, chest tube placement, and re-laparotomy within 30 days after the index operation or during patients' initial hospital stay
Assessment of additional oncological and perioperative outcomes: Kind of invasive re-interventions | 30 days after surgery
  Invasive re-interventions such as placement of interventional drains, Endoscopic retrograde cholangiopancreatography (ERCP) with stent placement, chest tube placement, and re-laparotomy within 30 days after the index operation or during patients' initial hospital stay
Assessment of additional oncological and perioperative outcomes: Number of patients with positive resection margins | During surgery
  Detection of tumor at the resection margin will be counted as positive resection margin
Assessment of additional oncological and perioperative outcomes: Frequency of Overall survival (OS) | 24 month
  The overall survival of all patients is assessed between operation date to date of death of any cause
Assessment of additional oncological and perioperative outcomes: Frequency of cancer-specific survival (CSS) | 24 months
  The cancer-specific survival of all patients is assessed between operation date to date of death of colorectal cancer
Assessment of additional oncological and perioperative outcomes: Frequency of disease-free survival (DFS) | 24 month
  The disease-free survival of all patients is assessed from operation date to the date of either progressive or recurrent disease, or death of any cause
Assessment of additional oncological and perioperative outcomes: Administration of adjuvant therapy [y/n] | 24 month
  Adjuvant therapy is not recommended. However, the decision for adjuvant therapy is left at discretion of the local oncologist. The administration of adjuvant therapy and kind of chemotherapy protocols used will be documented for both groups.
Assessment of additional oncological and perioperative outcomes: Frequency of oncological Re-interventions [y/n] | 24 month
  Frequency of interventions for treatment of intra- and/or extrahepatic disease recurrence will be documented. These interventions include: Chemotherapy, Surgical resection, Local ablation (e.g. radiofrequency or microwave ablation, stereotactic irradiation), Selective internal radiotherapy (SIRT), other
Assessment of additional oncological and perioperative outcomes: Kind of oncological Re-interventions [y/n] | 24 month
  Kind of interventions for treatment of intra- and/or extrahepatic disease recurrence will be documented. These interventions include: Chemotherapy, Surgical resection, Local ablation (e.g. radiofrequency or microwave ablation, stereotactic irradiation), Selective internal radiotherapy (SIRT), other
Assessment of additional oncological and perioperative outcomes: Assessment of "Quality of life" (QoL) | 12 month
  Quality of life is measured preoperatively and at 90 days (± 7 days) and 12 months (± 7 days) postoperatively using the EORTC QLQ-C30 questionnaire (European Organisation for Research and Treatment of Cancer; Questionnaire for the assessment of Quality of Life of Cancer patients with the module dedicated to colorectal liver metastases (EORTC QLQ-LMC21); the questionnaire assesses multi-item scales, each item scoring from 1 to 4, a high score represents a high level of symptomatology or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Weitz, Prof Dr med, Principal Investigator — Department of Gastrointestinal-, Thoracic and Vascular Surgery, University Hospital CGC; Nuh Rahbari, Prof Dr med, Principal Investigator — Allgemein- und Viszeralchirugie, University Hospital Ulm
Locations (37):
- Germany (37):
  - Department of Surgery at the University Medical Center Mannheim, Medical Faculty Mannheim, Heidelberg University, Mannheim, Baden-Wurttemberg
  - Department of Gastrointestinal-, Thoracic and Vascular Surgery University Hospital Carl Gustav Carus Technische Universität Dresden, Dresden, Saxony
  - Intestinal Center West Middle Franconia, ANregiomed Clinic Ansbach, Ansbach
  - Clinic for General, Vizeral and Transplant Surgery, Augsburg University Hospital, Augsburg
  - Department of General, Visceral and Vascular Surgery, Charité, University Medicine Berlin, Campus Benjamin Franklin Berlin, Berlin
  - Clinic and Polyclinic for General, Visceral, Thoracic and Vascular Surgery, University Hospital Bonn, Bonn
  - Surgical Clinic, Municipal Hospital Braunschweig gGmbH, Braunschweig
  - Cancer Center, Helios Amper-Hospital Dachau, Dachau
  - Surgical Clinic, Dortmund Hospital, Dortmund
  - Clinic for General and Visceral Surgery, Municipal Hospital Dresden, Dresden
  - Clinic for General, Visceral and Pediatric Surgery, University Hospital Düsseldorf, Düsseldorf
  - Surgical Clinic, University Hospital Erlangen, Erlangen
  - Clinic for General, Visceral and Transplant Surgery, University Hospital Frankfurt, Goethe University Frankfurt am Main, Frankfurt
  - Department for General and Visceral Surgery, Medical Center, University of Freiburg, Faculty of Medicine, University of Freiburg, Freiburg im Breisgau
  - JLU Gießen, Department for General, Visceral, Thoracic and Transplant Surgery, Giessen
  - Clinic for General, Visceral and Pediatric Surgery, University Medical Center Göttingen, Georg-August-University, Göttingen
  - Clinic and Polyclinic for General Surgery, Department of Gastrointestinal, Thoracic and Vascular Surgery, University Greifswald, University Hospital Greifswald, Greifswald
  - University Hospital and Polyclinic for Visceral, Vascular and Endocrine Surgery, University Hospital Halle (Saale), Halle
  - Center for Surgical Medicine - Clinic and Polyclinic for General, Visceral and Thoracic Surgery, University Hospital Hamburg-Eppendorf, Hamburg
  - Department of Liver, Bile Duct and Pancreas Surgery, University Department of surgery, Asklepios Klinik Barmbek, Hamburg
  - Clinic for General, Visceral and Minimally Invasive Surgery, KRH Clinic Siloah, Hannover, Hanover
  - Medizinische Hochschule Hannover, Department of General, Visceral and Transplant Surgery, Hanover
  - Department of General, Visceral and Transplantation Surgery, University of Heidelberg, Heidelberg
  - General Visceral and Vascular Surgery, Jena University Medical Center, Jena
  - Clinic for Surgery, University Hospital Schleswig-Holstein Lübeck Campus, Lübeck
  - University Department of General, Visceral, Vascular and Transplant Surgery, Faculty of Medicine, Otto von Guericke University Magdeburg, Magdeburg
  - Clinic for General, Visceral and Transplantation Surgery, University Medical Center of the Johannes Gutenberg-University Mainz, Mainz
  - Clinic for Visceral, Thoracic and Vascular Surgery, University Hospital Giessen and Marburg, Marburg
  - LMU Munich Hospital, Clinic for General, Visceral and Transplant Surgery, Munich
  - Department Hepato-Pancreato-Biliary Surgery, Barmherzige Brüder gGmbH of the Hospital Barmherzige Brüder Munich, München
  - Department of Surgery, University Hospital rechts der Isar, München
  - Clinic for General, Visceral and Transplant Surgery, University of Münster, Münster
  - University Hospital for General and Visceral Surgery, Oldenburg Hospital, Oldenburg
  - Department of General, Visceral and Transplant Surgery, University of Tübingen, Comprehensive Cancer Center, Tübingen
  - Clinic for General and Visceral Surgery, Ulm University Medical Center, Ulm
  - General and Visceral Surgery, Helios University Medical Center Wuppertal, University Witten/Herdecke, Wuppertal
  - Department for General, Visceral, Transplant, Vascular and Pediatric Surgery, Julius-Maximilian-University Würzburg, University Hospital Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: Undecided